CLINICAL TRIAL: NCT02173964
Title: Clinical Trial of Pinverin (Pinaverium Bromide) to Reduce Bowel Uptake of FDG in a Variety of Cancer Patients Who Undergo FDG PET/CT
Brief Title: Pinverin Application Trial to Reduce Bowel Uptake of FDG (Fluorodeoxyglucose)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Woo Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pin-2014-SNUBH
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: fluorodeoxyglucose; positron emission tomography; computed tomography; bowel; pinaverium bromide
MeSH Terms: conditions — Neoplasms | interventions — pinaverium; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pinaverium bromide (Experimental): pinaverium bromide 50 mg tablet per oral administration one time
  Interventions: Drug: pinaverium bromide
- water (Placebo Comparator): water ~100mL
  Interventions: Drug: water

INTERVENTIONS:
Drug: pinaverium bromide — pinverin 50 mg per oral single dose versus simple water ingestion
  Other Names: pinverin
  Arms: pinaverium bromide
Drug: water — same amount of water for pinverin administration
  Other Names: water~100mL
  Arms: water

SUMMARY:
1. Background

   1. PET/CT (positron emission tomography/computed tomography) using FDG (fluorodeoxyglucose) is widely used for evaluation of cancer patients.
   2. Bowel uptake of FDG is a serious problem that hampers the proper reading of PET/CT.
   3. There is no widely-accepted method to reduce the bowel FDG uptake.
2. Purpose

   1. To know whether pinverin (pinaverium bromide) application during PET/CT can reduce bowel uptake of FDG.
   2. Pinverin is a calcium-channel blocker that ameliorates the bowel contraction.
   3. Pinverin may be useful to reduce bowel FDG uptake by ameliorating the bowel contraction during PET/CT acquisition.
3. Method

   1. Intervention versus control: administration of single tablet of pinverin (50mg) perorally versus simple water (~100mL).
   2. Timing of administration: At the time of FDG injection. PET/CT images will be acquired 1hr post FDG injection.
4. Primary outcome

   1. SUV (standardized uptake value) difference between pinverin administered patient group versus control group.
   2. SUV (standardized uptake value) is calculated as: (decay corrected radioactivity in mCi/mL) x (body weight in g) / (injected radioactivity in mCi)

ELIGIBILITY:
Inclusion Criteria:

* Any cancer patients
* Candidate of positron emission tomography/computed tomography

Exclusion Criteria:

* Diabetes mellitus
* Inflammatory bowel disease
* Irritable bowel syndrome
* Peritoneal carcinomatosis
* Peritonitis
* Abdominal pain
* Diarrhea
* Medical test requiring bowel preparation within 1 month
* History of abdominal surgery
* Symptom or sign of colitis
* Pregnancy or lactation
* Hypersensitivity to pinaverium bromide
* Lactate intolerance
* Anit-depressant medication

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
SUV (standardized uptake value) | 1 hour after FDG (the radiopharmaceutical for PET/CT) injection
  SUV is the quantitative parameter of FDG uptake during PET/CT and represents the degree of relative FDG uptake in a specific lesion.
  SUV is calculated as: (decay-corrected radioactivity in mCi/mL) x (body weight in g) / (injected radioactivity in mCi). The unit of SUV is g/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Won Woo Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea